CLINICAL TRIAL: NCT03196739
Title: Feasibility of Virtual Reality Games Using Head-mounted Display on Patients With Brain Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Han Gil Seo, Clinical Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: VRfeasibility1.2
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2018-06-08 (Actual); Status verified 2018-03

CONDITIONS: Upper Extremity Dysfunction; Brain Diseases
MeSH Terms: conditions — Brain Diseases | interventions — Telerehabilitation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Virtual rehabilitation (Experimental): Upper limb rehabilitation using virtual reality with a head-mounted display (HTC Vive; HTC Co., New Taipei City, Taiwan)
  Interventions: Device: Virtual rehabilitation

INTERVENTIONS:
Device: Virtual rehabilitation — A total of 10 sessions were held for 30 minutes, 2 to 3 times a week for upper limb rehabilitation using immersive virtual reality under the assistance of an occupational therapist.

SUMMARY:
Because virtual reality can provide more enriched environment, repetitive goal-oriented tasks, and increased patients' interest and motivation, it is expected to stimulate neuroplasticity of injured brain and promote recovery in patients with brain disorders. On the other hand, immersive virtual reality using a head-mounted display has not yet been attempted in the rehabilitation of patients with brain disorders. In addition to the benefits of existing virtual reality or game rehabilitation, immersive virtual reality can further enhance brain plasticity, such as the effect of mirror therapy or action observation, through self-awareness of the body in the virtual space. The purpose of this study is to investigate the feasibility of applying the immersive virtual reality using a head-mounted display in patients with upper extremity dysfunction due to brain disorders.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper extremity dysfunction due to brain disorders (eg, stroke, traumatic brain injury, brain tumor, etc.)
* Patient who can move the upper limb against the gravity (MRC grade 3 or above in both shoulder and elbow flexion)
* Patient who can maintain stable sitting position
* Adults over 18 years old
* Patients who voluntarily agreed to participate in the study

Exclusion Criteria:

* A moderate-to-severe cognitive impairment score of 18 or less in Mini-Mental Status Examination (MMSE)
* Peripheral nerve injury, joint disease, other diseases of the upper extremity dysfunctions other than brain disorders
* Patients with a history of severe dizziness or epilepsy
* Patients with other medical illness that are difficult to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-06-06 (Actual)

PRIMARY OUTCOMES:
Change of Action Research Arm Test | at study completion, an average of 1 month
  19 items including grasp, grip, pinch, and gross arm movement

SECONDARY OUTCOMES:
Change of Box and Block Test | at study completion, an average of 1 month
  the number of blocks carried over the partition from one compartment to the other during the one-minute trial period
Change of Modified Barthel Index | at study completion, an average of 1 month
  Evaluation of activities of daily living
Time of participation | at study completion, an average of 1 month
  Total time of patient's participation in the study intervention
Patient's satisfaction | at study completion, an average of 1 month
  Evaluation of patient's satisfaction to the study intervention using a Likert scale
Patient's discomfort | at study completion, an average of 1 month
  Evaluation of patient's discomfort to the study intervention using a Likert

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Korea Workers' Compensation & Welfare Service Incheon Hospital, Incheon
  - Seoul National University Hospital, Seoul